CLINICAL TRIAL: NCT06955455
Title: Effectiveness of Ultrasound-Guided Corticosteroid and Bupivacaine Injections on Facial Nerve Function and Thickness in Acute Bell's Palsy: A Preliminary Trial
Brief Title: Ultrasound-Guided Corticosteroid and Bupivacaine for Facial Nerve Function and Thickness in Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University Hospital (Other)
Responsible Party: Principal Investigator, Ali Hammed, Dr, Tishreen University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N/2022-31; Tishreen University Hosital (Registry Identifier: Tsh-21)
Record Dates: First submitted 2025-04-18; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Bell's Palsy
MeSH Terms: interventions — Triamcinolone; Bupivacaine; Adrenal Cortex Hormones; Anesthetics, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-Guided Corticosteroid and Bupivacaine Injection (Experimental): Participants in this arm will receive a single, ultrasound-guided injection of 1 cc of 0.25% bupivacaine combined with 2 cc (20 mg) of triamcinolone (40 mg/mL). The injection is administered directly to the facial nerve (7th cranial nerve) approximately 1.5-2 cm distal to the stylomastoid foramen, in an inferior-anterior direction, under real-time ultrasound guidance. The goal is to reduce inflammation and accelerate recovery in patients with acute Bell's palsy.
  Interventions: Drug: Triamcinolone and Bupivacaine Injection

INTERVENTIONS:
Drug: Triamcinolone and Bupivacaine Injection — A single injection consisting of 1 cc of 0.25% bupivacaine mixed with 2 cc (20 mg) of triamcinolone (40 mg/mL) is administered under ultrasound guidance. The injection targets the extratemporal portion of the facial nerve approximately 1.5-2 cm distal to the stylomastoid foramen in an inferior and anterior direction. The intervention is designed to reduce inflammation and pain, potentially accelerating facial nerve recovery in acute Bell's palsy.
  Other Names: Corticosteroid and local anesthetic injection

SUMMARY:
This prospective, single-arm clinical study aims to evaluate the effects of a one-time, ultrasound-guided injection of corticosteroid (triamcinolone) combined with local anesthetic (bupivacaine) into the facial nerve in patients with acute Bell's palsy. The injection is administered approximately 1.5-2 cm after the nerve exits the stylomastoid foramen, with precise targeting using ultrasound imaging.

A total of 40 adult participants diagnosed within 72 hours of symptom onset will be enrolled. The primary outcome is improvement in facial nerve function, assessed using the House-Brackmann Facial Nerve Grading System at day 7, day 15, and 3 months post-injection. Secondary outcomes include changes in facial nerve thickness measured by ultrasound before and one week after the procedure.

This is the first clinical trial to directly evaluate targeted facial nerve injection as a potential treatment approach in Bell's palsy.

ELIGIBILITY:
Inclusion Criteria

Age between 18 and 70 years

Diagnosis of acute Bell's palsy within the past 72 hours

House-Brackmann Grade III or higher

Willing and able to give informed consent

Able to attend all follow-up assessments

Exclusion Criteria:

History of chronic facial nerve disorders

Known allergies to corticosteroids or local anesthetics

Coagulopathy or current use of anticoagulant therapy

MRI or CT findings indicating alternative causes of facial nerve palsy (e.g., tumor, stroke, MS)

Pregnancy or breastfeeding

Participation in another interventional clinical trial

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Improvement in facial nerve function using the House-Brackmann grading scale | 7 day, 15 days, and 3 months post-injection
  Facial nerve function will be assessed using the House-Brackmann Facial Nerve Grading System, a standardized clinical scale for measuring the severity of facial paralysis. Participants will be evaluated at three time points: 7 day, 15 days, and 3 months after injection. A reduction in grade indicates improvement in nerve function. This outcome will determine whether ultrasound-guided corticosteroid and bupivacaine injection accelerates recovery in acute Bell's palsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen University Hospital, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided